CLINICAL TRIAL: NCT00285662
Title: Intermittent Preventive Treatment (IPTi) for the Prevention of Malaria and Anaemia in PNG Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Papua New Guinea Institute of Medical Research (Other Government)
Collaborators: University of Melbourne (Other); Case Western Reserve University (Other)
Responsible Party: Prof Peter Siba, PNG Institute of Medical Research
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IPTi219
Record Dates: First submitted 2006-02-01; First posted 2006-02-02 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Malaria; Anemia
Keywords: IPTi; Malaria; Anemia; Prevention; Infant; Artesunate; SP; Amodiaquine; Papua New Guinea
MeSH Terms: conditions — Malaria; Anemia | interventions — Amodiaquine; fanasil, pyrimethamine drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): 1 day Sulfadoxine/Pyrimethamine + 3 days Amodiaquine
  Interventions: Drug: Amodiaquine/sulphadoxine-pyrimethamine, Artesunate/sulphadoxine-pyrimethamine or placebo
- 2 (Active Comparator): 1 day of Sulfadoxine/Pyrimthamine and 3 days of Artesunate
  Interventions: Drug: Amodiaquine/sulphadoxine-pyrimethamine, Artesunate/sulphadoxine-pyrimethamine or placebo
- 3 (Placebo Comparator): children of this gorup will receive only placebo dugs
  Interventions: Drug: Amodiaquine/sulphadoxine-pyrimethamine, Artesunate/sulphadoxine-pyrimethamine or placebo

INTERVENTIONS:
Drug: Amodiaquine/sulphadoxine-pyrimethamine, Artesunate/sulphadoxine-pyrimethamine or placebo — Children will get 25mg/1.25mg/kg of SP as a single dose, 4 mg/kg for 3 days of Artesunate and 10 mg/kg for 3 days of Amodiaquine in their respective arms

SUMMARY:
In malaria-endemic areas, young children have an especially high risk of malaria morbidity and mortality. Malaria is estimated to cause up to 2 million deaths and 500 million clinical episodes in Africa alone. The bulk of disease in Africa and severe disease and deaths globally is due to P. falciparum. However, P. vivax is also responsible for a substantial disease burden in endemic regions outside Africa, where P. vivax may account for more than half of all malaria cases. Efforts to reduce this unacceptably high disease burden are hampered by the limited availability of affordable interventions. Following the cessation of large-scale vector control in highly endemic areas, malaria control efforts have centred on early diagnosis and treatment of clinical cases and reducing exposure through the use of insecticide-treated nets (ITNs). While ITNs have been shown to significantly reduce the burden of malaria additional effective interventions are urgently needed.

Several trials have shown that chemoprophylaxis given to children at weekly or fortnightly intervals reduces morbidity from malaria in a number of different settings and populations.

An alternative approach has been to use intermittent preventive therapy (IPT) involving the administration of a full therapeutic dose of antimalarials at regular intervals. This is logistically easier to deliver, and is less costly, and may reduce problems of promoting drug resistance associated with regular chemoprophylaxis. Intermittent administration of sulphadoxine-pyrimethamine (SP) during antenatal clinic visits was shown to be highly effective in reducing malaria and anaemia in pregnant women and improving infant birth weights. IPT in pregnancy (IPTp) is now recommended by WHO for endemic regions of Africa.

DETAILED DESCRIPTION:
Intermittent preventive treatment in infancy (IPTi) is one of the most promising recent interventions to reduce the devastating impact of malaria in early childhood. Although two African studies have provided the proof of principle, further studies are needed to address several key issues. IPTi needs additional evaluation in a variety of settings and populations, alternative drugs and treatment schedules need to be tested and the long-term effect of IPTi on risk of malaria illness through early childhood needs to be clarified.

Many of these issues are currently being addressed in a series of studies conducted under the auspice of the IPTi Consortium. However, all these studies are based in sub-Saharan Africa and are thus almost exclusively concerned with the potential of IPTi to prevent P. falciparum malaria.

In order to determine whether IPTi is also an effective intervention in areas where there is a high prevalence of non-falciparum infections, further studies outside Africa are urgently needed. In addition, although initial IPTi studies have not shown a rebound in malaria morbidity following the intervention, the influence of IPTi on the acquisition of functional malaria immunity needs further investigation.

This proposal brings together investigators, experience, and resources to conduct a clinical trial of IPTi complemented by careful epidemiologic and laboratory investigations in two highly endemic areas of Papua New Guinea, where infections with all 4 human Plasmodium species are common. The studies will be based at the PNG Institute for Medical Research, which has excellent infrastructure and a strong history of malaria research and community-based studies

ELIGIBILITY:
Inclusion Criteria:

* 3 months old living in the aera for the next 2 years, exlusive use of the study health facilities

Exclusion Criteria:

* Known chronic illness, e.g. TB, diabetes, renal failure severe malnutrition (weight-for-age (WAZ) < 60% percentile) severe anaemia (Hb < 5 g/dl), or permanent disability, that prevents or impedes study participation

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1100 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of symptomatic malaria (due to any Plasmodium species) from 3 - 15 months of age | 15 months
Incidence of symptomatic P. falciparum malaria from 3 - 15 months of age | 15 months
Incidence of symptomatic P. vivax malaria from 3-15 months of age | !5 months

SECONDARY OUTCOMES:
Incidence of moderate-to-severe (Hb < 8 g/dl) and severe anaemia (Hb<5 g/dl) from 3 - 15 months of age | 15 months
Mean haemoglobin concentration and prevalence of moderate-to-severe anaemia (Hb < 8 g/dl) at 15 months of age | 15 months of age
Prevalence and density of malaria parasitemia at 15 months of age | 15 months
Prevalence of splenomegaly at 15 months of age | 15 months
Incidence of symptomatic malaria from 15 - 27 months of age | 27 months
9. Incidence of (symptomatic) moderate-to-severe (Hb < 8 g/dl) and severe anaemia (Hb<5 g/dl) from 15 - 27 months of age | 27 months
10. Mean haemoglobin levels and prevalence of moderate-to-severe (Hb < 8 g/dl) or severe anaemia at 27 months of age | 27 months
11. Prevalence and density of malaria parasitemia at 27 months of age | 27 months
12. Prevalence of splenomegaly at 27 months of age. | 27 months

CONTACTS AND LOCATIONS:
Overall Officials: Ivo Mueller, PhD, Principal Investigator — Papua New Guinea Institute of Medical Research; John Reeder, Prof, Principal Investigator — Papua New Guinea Institute of Medical Research
Locations (1):
- Papua New Guinea Institute of Medical Research, Goroka, Papua New Guinea

REFERENCES:
- [Derived] Senn N, Rarau P, Manong D, Salib M, Siba P, Reeder JC, Rogerson SJ, Genton B, Mueller I. Effectiveness of artemether/lumefantrine for the treatment of uncomplicated Plasmodium vivax and P. falciparum malaria in young children in Papua New Guinea. Clin Infect Dis. 2013 May;56(10):1413-20. doi: 10.1093/cid/cit068. Epub 2013 Feb 12. PMID 23403171
- [Derived] Senn N, Rarau P, Stanisic DI, Robinson L, Barnadas C, Manong D, Salib M, Iga J, Tarongka N, Ley S, Rosanas-Urgell A, Aponte JJ, Zimmerman PA, Beeson JG, Schofield L, Siba P, Rogerson SJ, Reeder JC, Mueller I. Intermittent preventive treatment for malaria in Papua New Guinean infants exposed to Plasmodium falciparum and P. vivax: a randomized controlled trial. PLoS Med. 2012;9(3):e1001195. doi: 10.1371/journal.pmed.1001195. Epub 2012 Mar 27. PMID 22479155
- [Derived] Senn N, Rarau P, Manong D, Salib M, Siba P, Robinson LJ, Reeder J, Rogerson S, Mueller I, Genton B. Rapid diagnostic test-based management of malaria: an effectiveness study in Papua New Guinean infants with Plasmodium falciparum and Plasmodium vivax malaria. Clin Infect Dis. 2012 Mar 1;54(5):644-51. doi: 10.1093/cid/cir901. Epub 2011 Dec 23. PMID 22198787